CLINICAL TRIAL: NCT05904964
Title: Disitamab Vedotin or Endocrine Therapy for Patients With Metastatic Breast Cancer With Hormone Receptor-positive and HER2-low-expression
Brief Title: Disitamab Vedotin (RC48) in Hormone Receptor Positive, HER2-low Metastatic Breast Cancer (the Rosy Trial)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Wang, Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-208-01
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: HR Positive/HER2 Low Expression Metastatic Breast Cancer
Keywords: HR positive; HRE2 low expression; metastatic breast cancer; ADC
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to disitamab vedotin or endocrine therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disitamab Vedotin (Experimental): Disitamab Vedotin, 2mg/kg, every 2 weeks
  Interventions: Drug: Disitamab vedotin
- Endocrine therapy (Active Comparator): Doctors choose endocrine therapy independently
  Interventions: Other: Endocrine therapy

INTERVENTIONS:
Drug: Disitamab vedotin — Disitamab Vedotin 2mg/kg was injected every 2 weeks,
  Other Names: RC48
  Arms: Disitamab Vedotin
Other: Endocrine therapy — Doctors choose endocrine therapy independently
  Arms: Endocrine therapy

SUMMARY:
Hormone receptor positive, HER2-low expression metastatic breast cancer is the main type of breast cancer, accounting for about 50% - 60%. However, this type of patients lack ideal therapeutic drugs after the failure of first-line standard endocrine therapy, and the median overall survival time is only 30 months. Therefore, finding more efficient and safe therapeutic drugs for these patients has become a big clinical challenge at present. Disitamab Vedotin (DV), as a new class I Antibody-Drug Conjugates drug, can achieve high efficiency and precise tumor killing effect with low toxicity. According to previous study with same sample size, DV also showed good efficacy in metastatic breast cancer with Hormone receptor positive and HER2- low expression as a posterior line treatment.Therefore, we intend to explore the efficacy and safety of DV in the treatment of HER2-low expressioin /Hormone receptor positive metastatic breast cancer patients with endocrine resistance through a scientifically designed, randomized, phase III clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (aged 18-70 years, including 18 and 70 years) with metastatic breast cancer confirmed by pathology or imaging are not suitable for surgical resection or radiotherapy for the purpose of cure;
2. Pathological examination confirmed that ER and / or PR were positive, and HER-2 was low expression (ER expression: immunohistochemical staining of tumor cells ≥ 10%; PR expression: immunohistochemical staining of tumor cells ≥ 10%; HER2-low: immunohistochemical staining of 2 + and FISH is not expanded, IHC 1 +);
3. Patients who have received endocrine therapy ;
4. According to the efficacy evaluation criteria for solid tumors (RECIST) version 1.1, there is at least one evaluable target lesion or only osteolytic bone metastasis;
5. Patients with stable brain metastasis or asymptomatic brain metastasis;
6. ECOG physical condition score ≤ 2 points, and the estimated survival time is not less than 3 months;
7. Prior treatment-related toxicity must be relieved to ≤ 1 degree (according to NCI CTCAE 5.0) before enrollment (except for hair loss or other toxicity that is considered as no risk to the safety of patients according to the judgment of the researcher);
8. Adequate bone marrow functional reserve: a. WBC ≥ 3.0 × 10 ^ 9 ／ L, b. Neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 ／ L, c. Platelet count (PLT) ≥ 70 × 10^9／L;
9. Liver, kidney and heart function tests were basically normal within one week before enrollment (based on the normal values of laboratories in each research center): A. total bilirubin (TBIL) ≤ 1.5 × upper limit of normal value (ULN), B. alanine aminotransferase (ALT / AST) ≤ 2.5 × ULN (liver metastasis patients ≤ 5xuln), C. serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 60 ml / min; d. left ventricular ejection fraction (LVEF) ≥ 55%, e. QTcF(Fridericia correction) ≤ 470 ms;
10. Patients understand the research process, voluntarily participate in the research, and sign the informed consent form.

Exclusion Criteria:

1. Patients who had received chemotherapy, radiotherapy, immunotherapy, and endocrine therapy for breast cancer within 2 weeks before enrollment.;
2. Patients who had performed major surgery within 2 weeks before enrollment.
3. Severe heart disease or discomfort within 12 months, including, but not limited to, the following: unstable angina pectoris, myocardial infarction, cerebral hemorrhage and cerebral infarction (except for silent lacunar cerebral infarction without treatment);
4. Have active autoimmune diseases (such as corticosteroids or immunosuppressive drugs) requiring systemic treatment in the past 2 years, excluding those with adrenal insufficiency requiring corticosteroid replacement therapy;
5. Have a clear history of neurological or mental disorders, including epilepsy or dementia;
6. According to the judgment of the researchers, there are some accompanying diseases that seriously endanger the safety of patients or affect patients to complete the study.
7. Those who have been known to have allergic history to Disitamab Vedotin or similar drugs;
8. According to the estimation of the investigator , the patient's compliance with the clinical study is insufficient or the researcher believes that there are other factors that are not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 24 months
  The interval from the date of randomization to the first imaging confirmed progression of disease or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
  The time interval from the date of randomization to death due to any cause.
Objective response rate (ORR) | 12 months
  According to recist1.1 standard, the proportion of patients whose best remission was CR or PR accounted for the total number of evaluable patients.
Disease Control Rate (DCR) | 12 months
  According to recist1.1 standard, the proportion of patients whose best remission was CR or PR or SD accounted for the total number of evaluable patients.
Clinical Benefit Rate (CBR) | 12 months
  According to recist1.1 standard, the proportion of patients whose best remission was CR or PR or SD ≥ 24 weeks accounted for the total number of evaluable patients.
Quality of life assessed by EORTC-C30 | 12 months
  Quality of life will be collected using the following questionnaire: EORTC-C30
Psychological condition assessed by GAD-7 | 12 months
Pittsburgh Sleep Scale | 12 months
Incidence of adverse events(AE) | from the date of enrollment to one year
  From the date of enrollment to one year, the incidence of adverse events in the fulvestrant combined with pyrotinib group was compared with that of capecitabine combined with pyrotinib group.
Biomarkers and treatment sensitivity analysis | 12 months
  Cox univariate and multivariate analysis will be used to explore the correlation between endocrine and HER2 pathway related biomarkers and treatment sensitivity（The biomarkers to be analyzed included 324 tumor related genes included in the FoundationOne CDx, and ER/PR/HER2/ki67 in IHC）

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (3):
- China (3):
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital， Shantou University Medical College, Shantou, Guangdong
  - Hainan Qionghai People's Hospital, Qionghai, Hainan

IPD SHARING:
Plan to Share IPD: No
Because the data involves the patient's personal information, it is temporarily decided that we will not disclose the individual participant data.

REFERENCES:
- [Background] Koleva-Kolarova RG, Oktora MP, Robijn AL, Greuter MJW, Reyners AKL, Buskens E, de Bock GH. Increased life expectancy as a result of non-hormonal targeted therapies for HER2 or hormone receptor positive metastatic breast cancer: A systematic review and meta-analysis. Cancer Treat Rev. 2017 Apr;55:16-25. doi: 10.1016/j.ctrv.2017.01.001. Epub 2017 Feb 20. PMID 28288388
- [Background] Mendes D, Alves C, Afonso N, Cardoso F, Passos-Coelho JL, Costa L, Andrade S, Batel-Marques F. The benefit of HER2-targeted therapies on overall survival of patients with metastatic HER2-positive breast cancer--a systematic review. Breast Cancer Res. 2015 Nov 17;17:140. doi: 10.1186/s13058-015-0648-2. PMID 26578067
- [Background] Wolff AC, Hammond MEH, Allison KH, Harvey BE, Mangu PB, Bartlett JMS, Bilous M, Ellis IO, Fitzgibbons P, Hanna W, Jenkins RB, Press MF, Spears PA, Vance GH, Viale G, McShane LM, Dowsett M. Human Epidermal Growth Factor Receptor 2 Testing in Breast Cancer: American Society of Clinical Oncology/College of American Pathologists Clinical Practice Guideline Focused Update. J Clin Oncol. 2018 Jul 10;36(20):2105-2122. doi: 10.1200/JCO.2018.77.8738. Epub 2018 May 30. PMID 29846122
- [Background] Giuliani S, Ciniselli CM, Leonardi E, Polla E, Decarli N, Luchini C, Cantaloni C, Gasperetti F, Cazzolli D, Berlanda G, Bernardi D, Pellegrini M, Triolo R, Ferro A, Verderio P, Barbareschi M. In a cohort of breast cancer screened patients the proportion of HER2 positive cases is lower than that earlier reported and pathological characteristics differ between HER2 3+ and HER2 2+/Her2 amplified cases. Virchows Arch. 2016 Jul;469(1):45-50. doi: 10.1007/s00428-016-1940-y. Epub 2016 Apr 21. PMID 27097809
- [Background] Schalper KA, Kumar S, Hui P, Rimm DL, Gershkovich P. A retrospective population-based comparison of HER2 immunohistochemistry and fluorescence in situ hybridization in breast carcinomas: impact of 2007 American Society of Clinical Oncology/College of American Pathologists criteria. Arch Pathol Lab Med. 2014 Feb;138(2):213-9. doi: 10.5858/arpa.2012-0617-OA. Epub 2013 Oct 28. PMID 24164555
- [Background] Modi S, Park H, Murthy RK, Iwata H, Tamura K, Tsurutani J, Moreno-Aspitia A, Doi T, Sagara Y, Redfern C, Krop IE, Lee C, Fujisaki Y, Sugihara M, Zhang L, Shahidi J, Takahashi S. Antitumor Activity and Safety of Trastuzumab Deruxtecan in Patients With HER2-Low-Expressing Advanced Breast Cancer: Results From a Phase Ib Study. J Clin Oncol. 2020 Jun 10;38(17):1887-1896. doi: 10.1200/JCO.19.02318. Epub 2020 Feb 14. PMID 32058843
- [Background] Yao X, Jiang J, Wang X, Huang C, Li D, Xie K, Xu Q, Li H, Li Z, Lou L, Fang J. A novel humanized anti-HER2 antibody conjugated with MMAE exerts potent anti-tumor activity. Breast Cancer Res Treat. 2015 Aug;153(1):123-33. doi: 10.1007/s10549-015-3503-3. Epub 2015 Aug 8. PMID 26253944
- [Background] Ocana A, Amir E, Pandiella A. HER2 heterogeneity and resistance to anti-HER2 antibody-drug conjugates. Breast Cancer Res. 2020 Jan 31;22(1):15. doi: 10.1186/s13058-020-1252-7. PMID 32005279
- [Background] Rios-Doria J, Harper J, Rothstein R, Wetzel L, Chesebrough J, Marrero A, Chen C, Strout P, Mulgrew K, McGlinchey K, Fleming R, Bezabeh B, Meekin J, Stewart D, Kennedy M, Martin P, Buchanan A, Dimasi N, Michelotti E, Hollingsworth R. Antibody-Drug Conjugates Bearing Pyrrolobenzodiazepine or Tubulysin Payloads Are Immunomodulatory and Synergize with Multiple Immunotherapies. Cancer Res. 2017 May 15;77(10):2686-2698. doi: 10.1158/0008-5472.CAN-16-2854. Epub 2017 Mar 10. PMID 28283653
- See also: NCCN Clinical Practical Guidelines in Oncology: Breast Cancer, Version 3.2021. — https://www.nccn.org/professionals/physician_gls/default.aspx